CLINICAL TRIAL: NCT01555489
Title: Phase II, Open Label Study of Intravenous Ascorbic Acid in Combination With Gemcitabine and Erlotinib in the Treatment of Metastatic Pancreatic Cancer
Brief Title: Assessing the Efficacy and Safety of IV Vitamin C in Combination With Standard Chemotherapy for Pancreatic Ca
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11D.365; JT 2181 (Other: JeffTrial Number)
Record Dates: First submitted 2012-02-22; First posted 2012-03-15 (Estimated); Results first posted 2018-08-28 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Stage IV Pancreatic Cancer
Keywords: Pancreatic Neoplasms; Pancreatic Cancer cells; Digestive System Neoplasms; Neoplasms by Site; Neoplasms; Endocrine Gland Neoplasms; Digestive System Diseases; Pancreatic Diseases; Endocrine System Diseases; Ascorbic Acid; Gemcitabine Vitamins; Vitamin C; Antioxidants; Molecular Mechanisms of Pharmacological Action; Pharmacologic Actions; Protective Agents; Physiological Effects of Drugs; Micronutrients; Growth Substances; Erlotinib; Integrative Medicine; Alternative Medicine; Complementary Medicine
MeSH Terms: conditions — Pancreatic Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Neoplasms; Endocrine Gland Neoplasms; Digestive System Diseases; Pancreatic Diseases; Endocrine System Diseases | interventions — Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ascorbic Acid, Gemcitabine & Erlotinib (Experimental): Ascorbic Acid (50-100g, 3x weekly) Standard Chemotherapy of Gemcitabine and Erlotinib for Pancreatic Cancer
  Interventions: Drug: Ascorbic Acid

INTERVENTIONS:
Drug: Ascorbic Acid — 3x per week
  Other Names: Vitamin C; Ascorbate

SUMMARY:
The investigators recently completed a phase I study of intravenous ascorbic acid (IV AA) plus standard chemotherapy (gemcitabine and erlotinib) in patients with metastatic pancreatic cancer. The investigators determined that the target ceiling dosage of 100 grams of ascorbic acid is safe when given with the chemotherapy. This Phase II trial is an initial test of efficacy of the 100 gram dose of ascorbic acid, which will be given with the same standard chemotherapy. This open label study will recruit up to 35 subjects with metastatic pancreatic cancer who will receive ascorbic acid combined with gemcitabine and erlotinib as front-line treatment. The phase I data suggests that ascorbic acid when given in combination with gemcitabine and erlotinib may result in some tumor response, and the goal of this study is to better evaluate the response and confirm initial safety data

DETAILED DESCRIPTION:
Intravenous high dose ascorbic acid is a widely used alternative cancer treatment. Patients will receive standard care gemcitabine/erlotinib for treatment of their metastatic pancreatic adenocarcinoma. They will be closely monitored for disease response/ progression. If vitamin C has a beneficial effect on tumour cells, patients may experience a regression of tumor or tumor markers. Additional benefits include scans at no charge to the patient. This study requires several days of treatment per week and treatments are given in two different locations. The intravenous vitamin C treatments are given 3 times per week, these are given every week for an initial cycle of 15 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Males and females of age ≥ 18
* Histologically or cytologically confirmed pancreatic adenocarcinoma that has metastatic disease measurable by CT, MRI, or PET
* Subjects with unresectable pancreatic cancer who have had surgery (exploratory laparotomy, biliary, gastrointestinal bypass) are eligible, if the subject has fully recovered from surgery and ≥ 14 days has passed since the operation. Patients with history of pancreatoduodenectomy are eligible provided that there is radiographically documented disease recurrence.
* ECOG performance status 0-2
* Laboratory values that would not prevent the patient from receiving chemotherapy as determined by the PI or study oncologist
* G6PD status ≥ lower limit of normal
* Serum creatinine ≤ 2.0 mg/dL

Exclusion Criteria:

* Islet cell or acinar cell carcinoma or cystadenocarcinoma
* History or known presence of central nervous system (CNS) metastases
* History of another primary cancer, except:
* Curatively treated cervical carcinoma in situ, or
* Curatively resected non-melanomatous skin cancer, or
* Other primary solid tumor curatively treated with no known active disease present and no treatment administered for ≥ 3 years prior to enrollment
* Other concurrent anticancer chemotherapy
* Prior radiotherapy ≤ 14 days, or if subjects have not recovered from radiotherapy
* Uncontrolled seizure disorder or other serious neurological diseases
* Any co-morbid disease that would increase risk of toxicity as determined by PI
* Only locally advanced disease
* Prior treatment with gemcitabine (for metastatic pancreatic cancer)
* Subjects requiring chronic use of immunosuppressive agents (eg, methotrexate, cyclosporine, corticosteroids)
* Recent infection requiring a course of systemic anti-infection that was completed ≤ 14 days prior to enrollment (exception can be made at the judgment of the PI for oral treatment of an uncomplicated urinary tract infection ([UTI])
* History of any medical or psychiatric condition or addictive disorder, or laboratory abnormality that, in the opinion of the PI, may increase the risks associated with study participation or study drug administration or may interfere with the conduct of the study or interpretation of study requirements
* Subject unwilling or unable to comply with study requirements
* Subject who is pregnant or breast feeding
* Known positive test(s) for human immunodeficiency virus infection, hepatitis C virus, chronic active hepatitis B infection
* Documented history of alcohol, cocaine or intravenous drug abuse ≤ 6 months of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A Monti, MD, Principal Investigator — Thomas Jefferson University; Edith P Mitchell, MD, Study Chair — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Monti DA, Mitchell E, Bazzan AJ, Littman S, Zabrecky G, Yeo CJ, Pillai MV, Newberg AB, Deshmukh S, Levine M. Phase I evaluation of intravenous ascorbic acid in combination with gemcitabine and erlotinib in patients with metastatic pancreatic cancer. PLoS One. 2012;7(1):e29794. doi: 10.1371/journal.pone.0029794. Epub 2012 Jan 17. PMID 22272248
- See also: Phase I results — http://www.plosone.org/article/info%3Adoi%2F10.1371%2Fjournal.pone.0029794

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ascorbic Acid, Gemcitabine & Erlotinib
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ascorbic Acid, Gemcitabine & Erlotinib
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Safety of Ascorbic Acid in Combination With Gemcitabine and Erlotinib for Stage IV Pancreatic Cancer
Description: Safety: to assess safety of IVAA in combination with gemcitabine and erlotinib by evaluating the number of adverse events and serious adverse events occurring among study participants.
Time Frame: 15 weeks
Population: The trial was closed due to lack of accrual. The standard of care treatment that was part of the study as initially written changed to a different chemotherapy regimen thus not enabling the team to enroll additional patients. The data were not collected.
Arm/Group | Ascorbic Acid, Gemcitabine & Erlotinib
Number analyzed (Participants) | 0

2. Secondary Outcome: Evaluate Quality of Life Using Functional Assessment of Cancer Therapy-General (FACT-G) Quality Assessment Instrument
Description: 1) To evaluate quality of life using Functional Assessment of Cancer Therapy-General (FACT-G) quality assessment instrument. The FACT-G questionnaire as well as the Patient Reported Outcomes Measurement Information System (PROMIS-29) will be used to assess quality-of-life longitudinally. Quality-of-life scores obtained from the FACT-G and PROMIS-29 will be summarized at multiple time points using means and standard deviations.
Time Frame: 15 weeks
Population: as for outcome 1
Arm/Group | Ascorbic Acid, Gemcitabine & Erlotinib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Ascorbic Acid, Gemcitabine & Erlotinib
All-Cause Mortality (participants affected / at risk) | 1/11
Serious Adverse Events (participants affected / at risk) | 1/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ascorbic Acid, Gemcitabine & Erlotinib (N=11)
Death (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ascorbic Acid, Gemcitabine & Erlotinib (N=11)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Low hemoglobin (Blood and lymphatic system disorders) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Infection with normal ANC (Immune system disorders) | 1 (1)
Low platelets (Blood and lymphatic system disorders) | 2 (3)
GI Obstruction (Gastrointestinal disorders) | 1 (1)
Increased creatinine (Blood and lymphatic system disorders) | 1 (1)
Nausea (General disorders) | 1 (1)
Low Potassium (Blood and lymphatic system disorders) | 1 (1)
Cardiac Infarction (Cardiac disorders) | 1 (1)
Sepsis (Immune system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes